CLINICAL TRIAL: NCT01210508
Title: A Prospective Analysis of the Tokuhashi Score and Its Effectiveness in Guiding Treatment and Predicting Survival in Patients With Metastases Spread to the Spine
Brief Title: Analysis of Tokuhashi Score
Status: Terminated | Type: Observational
Why Stopped: low enrollment
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Cleveland Clinic Florida (Other)
Responsible Party: Principal Investigator, William Lavelle, Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: IRB 5797
Record Dates: First submitted 2010-01-26; First posted 2010-09-28 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2013-09

CONDITIONS: Cancer; Metastases
Keywords: Cancer patients with metastases to the spinal column
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
70% of all cancer patients develop some form of visceral (internal organs) or skeletal metastases (spread of disease). Approximately one third of cancer patients develop metastases to the spinal column. The prognosis once spinal metastases have been diagnosed and the most appropriate treatment still remains controversial. To date there is no one good diagnostic tool to predict survival and/or outcome after radiotherapy or surgical intervention.

Tokuhashi, et al, formulated and presented a preoperative scoring system to evaluate indications for surgery and predict outcome in patients with metastases to the spinal column. Six variables are measured to calculate this score: general medical condition, number of extraspinal metastases, number of vertebral metastases, status of metastases to the major internal organs, primary tumor type, and presence of a neurologic deficit. This scoring system has been gaining acceptance in literature. In 1998, Tokuhashi, et al, modified this scoring system by diversifying the tumor types into six categories. After a retrospective analysis Tokuhashi reported that patients with scores less than or equal to 8 will die of their disease within 6 months and those with scores of 12 or greater will survive an average of 12 months or more.

The purpose of this study is to determine 1) the Tokuhashi score's validity in predicting survival after developing spinal metastases, 2) the relationship of treatment on survival after detecting spinal metastases in relation to the Tokuhashi score. Patients will be enrolled into the study and followed prospectively for as long as possible regardless of intervention.

There will be three groups based on their Tokuhashi score, each group will require approximately 163 subjects statistically.

DETAILED DESCRIPTION:
all info is in brief summary

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with any form of spinal metastases, whether symptomatic or not, regardless of tumor biology, and seen by a physician in the Department of Orthopedic Surgery, will be asked to enter this trial.
* Must be a patient of our practice

Exclusion Criteria:

* There is no exclusion criteria

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen in the Orthopedic Spine office, that have been diagnosed with metastases to the spine.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine the Tokuhashi score's validity in predicting survival after developing spinal metastases | 24 months
  will follow subjects until death

SECONDARY OUTCOMES:
the relationship of treatment on survival after detecting spinal metastases in relation to the Tokuhashi score | 24 months
  will follow subjects until death

CONTACTS AND LOCATIONS:
Overall Officials: William F. Lavelle, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Upstate Orthopedic Bone and Joint Center, East Syracuse, New York, United States